CLINICAL TRIAL: NCT02967744
Title: BEVAR: Patientspecifik Behandling Ved Artrose - Et "Proof-of-concept"- Kvalitetssikringsstudie
Brief Title: NSAID Treatment of Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Kristian Kjær Petersen, assistant professor, Aalborg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: N-20140077
Record Dates: First submitted 2016-11-14; First posted 2016-11-18 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis,Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NSAID treatment (Experimental): 8 weeks of NSAID treatment
  Interventions: Drug: NSAID

INTERVENTIONS:
Drug: NSAID — NSAIDs are among the most common pain treatments for patients with osteoarthritis.

SUMMARY:
The study investigates associations between pre treatment pain intensity and central pain mechanisms on the effect of 8-week treatment of NSAIDs in patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Knee Ostoarthritis

Exclusion Criteria:

* Current ulcer diagnosed by endoscope
* Asthma or other allergic reaction to NSIADs
* Kidney disease
* Myocardial infarction within the last six months
* Severe hyper tension (systolic ≥180mmHg, diastolic ≥110mmHg)
* Severe thrombocytopenia (thrombocyst count <50x10^9/l)
* Insufficience lever or kidney function

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2016-01; Primary Completion 2018-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured on a 10cm visual analog scale | 8 weeks after treatment
  Patients will be asked to rate the pain intensity 8 weeks after treatment on a 10cm visual analog scale (0 indicating no pain, 10 indicating worst imaginable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sensory Motor Interaction, Aalborg University, Aalborg East, Denmark

REFERENCES:
- [Derived] Giordano R, Arendt-Nielsen L, Hertel E, Olesen AE, Petersen KK. Multifactorial Machine Learning Algorithm Integration of Pain Mechanisms Can Predict the Efficacy of 3-Week NSAID Plus Paracetamol in Patients With Painful Knee Osteoarthritis. Eur J Pain. 2025 Nov;29(10):e70140. doi: 10.1002/ejp.70140. PMID 41020650
- [Derived] Hertel E, Arendt-Nielsen L, Olesen AE, Andersen MS, Petersen KK. Quantitative sensory testing, psychological factors, and quality of life as predictors of current and future pain in patients with knee osteoarthritis. Pain. 2024 Aug 1;165(8):1719-1726. doi: 10.1097/j.pain.0000000000003194. Epub 2024 Feb 20. PMID 38381930